CLINICAL TRIAL: NCT06935877
Title: Comparison of the Efficacy of Combined Hyaluronic Acid and Triamcinolone Acetonide Injection and Hyaluronic Acid Alone Injection in Patients With Subdeltoid Bursitis
Brief Title: Additional Effect of Steroid on Hyaluronic Acid in Subdeltoid Bursitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, MD, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025SKHADR040
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Subdeltoid Bursitis of the Shoulder
MeSH Terms: interventions — Hyaluronic Acid; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): traditional rehabilitation programs
  Interventions: Drug: Hyaluronic acid injection; Drug: Triamcinolone Acetonide injection
- Control (Active Comparator): Hyaluronic acid injection
  Interventions: Drug: Hyaluronic acid injection

INTERVENTIONS:
Drug: Hyaluronic acid injection — traditional rehabilitation programs
  Other Names: Hyaluronic acid
Drug: Triamcinolone Acetonide injection — traditional rehabilitation programs
  Other Names: Triamcinolone Acetonide
  Arms: Intervention group

SUMMARY:
The study employs a double-blind, randomized clinical trial design with 60 patients diagnosed with subdeltoid bursitis. Participants are divided into two groups: the experimental group receives combined hyaluronic acid and Triamcinolone Acetonide injections, while the control group receives hyaluronic acid alone injection. All injections are guided by ultrasound. Assessments are conducted before treatment and at 1 week, 1 month, and 3 months post-treatment.

DETAILED DESCRIPTION:
Evaluation indicators include pain (measured by Visual Analog Scale for rest, activity, and sleep, and pain threshold via pressure algometer), function (assessed by Disabilities of the Arm, Shoulder, and Hand score and Shoulder Pain and Disability Index), quality of life (using the World Health Organization Quality of Life-BREF).

ELIGIBILITY:
Inclusion Criteria:

* - Unilateral shoulder pain within the past 3 months

Pain during joint movements such as abduction or internal rotation

At least one positive result from the following tests: Painful arc, Neer test, or Hawkins test

No shoulder injections received in the past 3 months

Willingness to receive injection treatment and undergo follow-up assessments at the following time points:

Immediate (1 week after injection)

Short-term (1 month after injection)

Mid-term (3 months after injection)

Avoid use of anti-inflammatory painkillers during the study period as much as possible; if intolerable pain occurs, acetaminophen (provided by the researcher) will be used to relieve symptoms

Exclusion Criteria:

* Presence of infectious disease, inflammation, rheumatoid arthritis, or fracture

History of malignancy

Previous shoulder surgery

Sensory deficits

Tendon rupture of the rotator cuff or biceps tendon

Neurological disorders causing hand weakness or affecting shoulder mobility (e.g., stroke, Parkinson's disease, brachial plexus injury, peripheral neuropathy)

Cognitive impairment preventing completion of questionnaires

Cervical radiculopathy

Diagnosed frozen shoulder (adhesive capsulitis)

Psychiatric disorders

Breastfeeding or pregnant women

Received shoulder injection within the past 3 months, including corticosteroids, hyaluronic acid, Platelet-rich plasma, or any prolotherapy solution

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index | Score change from baseline to 1 week, 1 months and 3 months of treatment, higher score, the better outcome
  A questionnaire to evaluate the severity of shoulder pain and disability in patients with shoulder problems; higher scores indicated more significant pain and disability.The score ranges from 0 to 100: 0 = no disability; 100 = most severe disability

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand | Score change from baseline to 1 week, 1 months and 3 months of treatment, higher score, the better outcome
  The questionnaire to measure physical function and symptoms in people with upper-limb disorders, including conditions affecting the shoulder, elbow, wrist, or hand. The score ranges from 0 to 100: 0 = no disability; 100 = most severe disability
Score change from baseline to 1 week, 1 months and 3 months of treatment, higher score, the better outcome | Score change from baseline to 1 week, 1 months and 3 months of treatment, higher score, the better outcome
  Range of motions of shoulder joint
World Health Organization Quality of Life | Score change from baseline to 1 week, 1 months and 3 months of treatment, higher score, the better outcome
  Assesses 4 key domains: Physical Health, Psychological , Social Relationships and Environment, score ranges 0-100, higher score indicates greater health
visual analog scale | Score change from baseline to 1 week, 1 months and 3 months of treatment, higher score, the better outcome
  Measuring subjective pain intensity, score ranges from 0 to 10 (or 0 to 100 mm, depending on format), the higher score indicates more severe symptom

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, Study Director — Shin Kong Wu Ho-Su Memorial Hospital

IPD SHARING:
Plan to Share IPD: No